CLINICAL TRIAL: NCT07140029
Title: Comparative Clinical Study of Intraocular Lens Injectors Lioli™, Pioli™, and Pioli™ Plus
Status: Recruiting | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PIOLI012022
Record Dates: First submitted 2025-03-21; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-03

CONDITIONS: Cataract; Lens Implantation, Intraocular
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- pioli™ rD: Participants receiving the pioli™ preloaded injector with the rD model, used for IOL powers < 25.5 diopters
- pioli™ Plus rD: Participants receiving the pioli™ Plus preloaded injector with the rD model, used for IOL powers < 25.5 diopters
- lioli™ <25.5D: Participants receiving the lioli™ manually loaded injector for IOL powers < 25.5 diopters
- pioli™ rC: Participants receiving the pioli™ preloaded injector with the rC model, used for IOL powers ≥ 25.5 diopters
- pioli™ Plus rC: Participants receiving the pioli™ Plus preloaded injector with the rC model, used for IOL powers ≥ 25.5 diopters
- lioli™ ≥25.5D: Participants receiving the lioli™ manually loaded injector for IOL powers ≥ 25.5 diopters

SUMMARY:
The goal of this observational study is to evaluate whether different intraocular lens (IOL) injectors affect surgical outcomes in patients aged 40 and older undergoing cataract surgery. The main questions it aims to answer are:

* Do different IOL injectors change the size of the corneal incision during surgery?
* Do the injectors lead to different rates of complications during or after surgery? Researchers will compare the use of three different IOL injectors: two preloaded models (pioli™ and pioli™ Plus) and one manually loaded model (lioli™), to see if the preloaded systems improve surgical results compared to the manual one.

Participants will:

* Undergo routine cataract surgery using one of the three injectors, randomly assigned.
* Have measurements taken before and after surgery (e.g., vision tests, corneal incision size).
* Be monitored for any side effects or complications during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Scheduled for cataract surgery using phacoemulsification technique
* Planned implantation of an Asqelio™ monofocal intraocular lens (IOL)
* Clear intraocular media, except for the presence of cataract (i.e., no other significant ocular opacities)

Exclusion Criteria:

* Preoperative corneal astigmatism > 1.0 diopter (D)
* Previous corneal surgery or history of ocular trauma
* Irregular cornea (e.g., keratoconus)
* Choroidal hemorrhage
* Microphthalmos
* Severe corneal dystrophy
* Uncontrolled or medically controlled glaucoma
* Clinically significant macular changes
* Severe concomitant ocular disease
* Cataract not related to aging
* Severe optic nerve atrophy
* Diabetic retinopathy
* Proliferative diabetic retinopathy
* Amblyopia
* Extremely shallow anterior chamber
* Severe chronic uveitis
* Pregnant or breastfeeding
* Rubella
* Mature or dense cataracts that prevent preoperative retinal examination
* History of retinal detachment
* Concurrent participation in another drug or medical device clinical study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 40 and older) scheduled for routine cataract surgery using phacoemulsification and implantation of an Asqelio™ monofocal intraocular lens. Participants must have clear intraocular media except for the presence of cataract and meet standard clinical criteria for lens implantation. Patients are recruited from a single ophthalmology center in Spain and are typical candidates for conventional cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Corneal Incision Size | Day of surgery (intraoperative)
  Measurement of the corneal incision before and after intraocular lens (IOL) insertion using each type of injector. Difference in incision size (in mm)
Incidence of Adverse Events | From surgical incision to end of surgery, assessed up to 120 minutes (intraoperative), and From end of surgery until postoperative day 30 (postoperative)
  Number and type of ocular and non-ocular adverse events (serious and non-serious) recorded from initiation of the intra-ocular lens (IOL) implantation, both intraoperative and early postoperative period (up to 30 days). Percentage of participants with any AE

SECONDARY OUTCOMES:
Procedure Duration | During surgery
  Time required to insert the IOL using each type of injector. Time in seconds (measured with a stopwatch)

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Hernández Martínez, MD, PhD, Principal Investigator — OftalVist Sevilla
Locations (1):
- Clínica OftalVist Sevilla, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No
The study does not include a plan to share individual participant data (IPD), as data will be anonymized and used solely for internal analysis and regulatory reporting